CLINICAL TRIAL: NCT03771898
Title: A Global, Multicenter, Single-arm, Matched External Control Study of Intrathecal SHP611 in Subjects With Late Infantile Metachromatic Leukodystrophy
Brief Title: A Study of Intrathecal SHP611 in Children With Metachromatic Leukodystrophy
Acronym: EMBOLDEN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP611-201; 2018-003291-12 (EudraCT Number); jRCT2041200086 (Registry Identifier: jRCT)
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Metachromatic Leukodystrophy (MLD)
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SHP611 (Experimental): Participants will receive 150 milligrams (mg) of SHP611 intrathecally (IT) via intrathecal drug delivery device (IDDD) or lumbar puncture (LP) once weekly for 106 weeks in six groups (Group A, B, C, D, E, and F) based on participant's age and motor dysfunction.
  Interventions: Drug: SHP611

INTERVENTIONS:
Drug: SHP611 — Participants will receive 150 mg of SHP611 IT via IDDD or LP once weekly for 106 weeks.
  Other Names: HGT-1110, TAK-611; recombinant human arylsulfatase A [rhASA]

SUMMARY:
The main aim of the study is to determine if SHP611 given by injection into the spinal fluid that surrounds the brain and spinal cord (intrathecal; IT) prolongs the time for children with Metachromatic Leukodystrophy (MLD) to retain the ability to move from place to place. Other aims of the study are to determine the effects of intrathecal administration of SHP611 on movement and speech functions and to learn how well SHP611 injected in the spinal fluid that surrounds the brain and spinal cord is tolerated.

Study participants will receive SHP611 for about 2 years with the possibility of an extended treatment period.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have a documented diagnosis of MLD (Groups A-F):

  1. Low ASA activity in leukocytes (compared to laboratory normal range).
  2. Elevated sulfatides in urine.
* The participant must have a gait disorder due to spastic ataxia or weakness attributable to MLD by the investigator and documented by a primary care physician or a specialist physician by 30 months of age (Groups A-C, and F), or be minimally symptomatic and greater than or equal to (> =) 6 to less than (<) 18 months of age (Group D) or be early symptomatic and > =12 to < 18 months of age (Group E). Participants in Group E must have neurological symptoms either documented by either a primary care physician or a specialist physician.
* The participant's age at the time of informed consent, must be: Group A: 18 to 48 months of age; Group B: 18 to 72 months of age; Group C: 18 to 72 months of age; Group D: >= 6 to < 18 months of age; Group E: > = 12 to < 18 months of age; Group F: 18 to 72 months of age.
* The participant's GMFC-MLD category at screening must be: Group A: GMFC-MLD category of 1 or 2; Group B: GMFC-MLD category of 3; Group C: GMFC-MLD category of 4; Group D: minimally symptomatic, >= 6 to < 18 months of age, with the same arylsulfatase (ASA) allelic constitution as an older sibling with confirmed late infantile or juvenile onset MLD; Group E: early symptomatic, >= 12 to < 18 months of age with a GMFC-MLD category of 1 or 2 with a history of achieving stable walking (defined as at least 1 month of independent walking); Group F: GMFC-MLD category of 5 or 6.
* The participant and his/her parent/representative(s) must have the ability to comply with the clinical protocol.
* Participant's parent or legally authorized representative(s) must provide written informed consent prior to performing any study-related activities. Study-related activities are any procedures that would not have been performed during normal management of the participant.

Exclusion Criteria:

* Multiple sulfatase disorder as determined by abnormal activity of another lysosomal sulfatase (based upon the reference laboratory's normal range) or a known genetic disorder other than MLD.
* History of bone marrow transplant (BMT), hematopoietic stem cell transplantation (HSCT), or gene therapy; or undergoes BMT, HSCT, or gene therapy: at any point during the study.
* Primary presentation of MLD was behavioral or cognitive symptoms (per investigator's clinical judgment); behavioral symptoms that are secondary to motor deficits (example [eg], tantrums in response to loss of motor skills) are not exclusionary.
* The participant has any known or suspected hypersensitivity to agents used for anesthesia or has history of difficult airway or potential for airway compromise.
* Any other medical condition or serious comorbid illness that in the opinion of the investigator would preclude participation in the study.
* Participants with laboratory, ECG or vital sign abnormalities reflecting intercurrent illness that may compromise their safety during the trial should not be enrolled. Abnormal laboratory, vital sign and ECG results at screening should be reviewed with the Takeda medical monitor.
* The participant is enrolled in another clinical study that involves use of any investigational product (drug or device) within 30 days or 5 half-lives (whichever is longer) prior to study enrollment or at any time during the study.
* The participant has had prior exposure to SHP611.
* The participants must weigh > 11 pound (lbs) (5 kilograms [kg]).
* The participant has a condition that is contraindicated as described in the SOPH-A-PORT Mini S IDDD Instructions for Use (IFU)

  1. The participant has had, or may have, an allergic reaction to the materials of construction.
  2. The participant has shown an intolerance to an implanted device.
  3. The participant's body size is too small to support the size of the SOPH-A-PORT Mini S Access Port.
  4. The participant's drug therapy requires substances known to be incompatible with the materials of construction.
  5. The participant has a known or suspected local or general infection.
  6. The participant is at risk of abnormal bleeding due to a medical condition or therapy.
  7. The participant has one or more spinal abnormalities that could complicate safe implantation or fixation.
  8. The participant has a functioning Cerebro spinal fluid(CSF) shunt device .

Matched External Control Participants for Group A from Global Leukodystrophy Initiative of Metachromatic Leukodystrophy (GLIA-MLD) The matched external control group must have data for at least baseline gross motor function evaluation. Selection of the external control participants from GLIA-MLD will follow a set of criteria as similar as possible to the inclusion criteria for Group A in the SHP611-201 study protocol.

A filtering process will be applied to select the external control participants from the GLIA-MLD database, by meeting all of the following 3 filtering criteria:

1. Filtering criterion 1: requiring documented diagnosis of MLD, based on

   * low arylsulfatase A (ASA) activity in leukocytes AND elevated sulfatides in urine. OR
   * biallelic variants in arylsulfatase A gene (ARSA) AND (either low ASA activity in leukocytes OR elevated sulfatides in urine).
2. Filtering criterion 2: requiring documented gait disorder. Participants will be considered qualifying if they present with a gait disorder before 2.5 years (30 months) of age and have a medical record reporting a gait abnormality including, but not limited to, the following terms: ataxia, spasticity, and hyper/hypotonia.
3. Filtering criterion 3: participants will be considered qualifying if they have at least 1 clinical encounter occurring between the age of 18 to 48 months with a GMFC-MLD category either 1 or 2.

Ages: 6 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2026-03-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (30):
- United States (11):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA, Torrance, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - New York University Langone Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Hospital Universitario Austral - PIN, Ciudad Autónoma Buenos Aires, Buenos Aires, Argentina
- UZ Antwerpen, Edegem, Belgium
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil
- Canada (4):
  - Stollery Children's Hospital University of Alberta, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- France (2):
  - Hôpital Bicêtre - Paris Sud, Le Kremlin-Bicêtre
  - CHU Lenval, Nice
- Germany (2):
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Tübingen, Tübingen
- Attikon University General Hospital, Chaïdári, Attica, Greece
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- IRCCS Ospedale Pediatrico Bambino Gesù - INCIPIT - PIN, Roma, Italy
- Kanazawa University Hospital, Kanazawa, Japan
- VU Medisch Centrum, Amsterdam, Netherlands
- Spain (2):
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Vall d'Hebrón, Barcelona
- Birmingham Children's Hospital NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd64db2bf003ab46e0b

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 19 investigational sites. A total of 36 participants were enrolled in this two-period study (primary treatment and extension periods) of which 35 received SHP611 or had intrathecal drug delivery device (IDDD) implanted. Data was reported till the primary treatment period. The study is still ongoing, additional data will be reported after the completion of the study. Study consisted of six groups (Group A,B,C,D, E, F) based on participant's age and motor dysfunction.
Pre-assignment Details: No participants were enrolled in Groups D and E, hence no data was collected or reported for these two groups. For efficacy analysis, Group A arm of current study was compared with matched external control group (33 participants) data from untreated metachromatic leukodystrophy (MLD) participants in the Global Leukodystrophy Initiative natural history study (GLIA-MLD), part of the Global Leukodystrophy Initiative Clinical Trials Network (GLIA-CTN, NCT03047369).
Groups:
- Group A, SHP611: Participants aged 18 to 48 months with Gross Motor Function Classification in Metachromatic Leukodystrophy (GMFC-MLD) Category of 1 or 2 received SHP611 150 milligrams (mg) intrathecally (IT) via IDDD or lumbar puncture (LP), once weekly for 106 weeks in primary treatment period. Participants who completed primary treatment period will be continued treatment in extension period up to Week 210 or beyond, until their parents/guardians decided to discontinue treatment; the sponsor discontinued the study; the participant discontinued from the study due to medical or safety concerns; or the product became commercially available in the participant's country of residence, whichever came first.
- Group B, SHP611: Participants aged 18 to 72 months with GMFC-MLD Category of 3 received SHP611 150 mg IT via IDDD or LP once weekly for 106 weeks in primary treatment period. Participants who completed primary treatment period will be continued treatment in extension period up to Week 210 or beyond, until their parents/guardians decided to discontinue treatment; the sponsor discontinued the study; the participant discontinued from the study due to medical or safety concerns; or the product became commercially available in the participant's country of residence, whichever came first.
- Group C, SHP611: Participants aged 18 to 72 months with GMFC-MLD Category of 4 received SHP611 150 mg IT via IDDD or LP once weekly for 106 weeks in primary treatment period. Participants who completed primary treatment period will be continued treatment in extension period up to Week 210 or beyond, until their parents/guardians decided to discontinue treatment; the sponsor discontinued the study; the participant discontinued from the study due to medical or safety concerns; or the product became commercially available in the participant's country of residence, whichever came first.
- Group F, SHP611: Participants aged 18 to 72 months with GMFC-MLD Category of 5 or 6 received SHP611 150 mg IT via IDDD or LP once weekly for 106 weeks in primary treatment period. Participants who completed primary treatment period will be continued treatment in extension period up to Week 210 or beyond, until their parents/guardians decided to discontinue treatment; the sponsor discontinued the study; the participant discontinued from the study due to medical or safety concerns; or the product became commercially available in the participant's country of residence, whichever came first.
- GLIA-MLD Matched External Control for Group A: Group A matched external control group of untreated MLD participants (who have received no investigational product or therapy) from the ongoing GLIA-MLD retrospective natural history study with exact matching GMFC-MLD score with Group A were selected. The GLIA-MLD natural history study database was used as source data for external control matching group participants for efficacy comparison.
Period: Overall Study
Arm/Group | Group A, SHP611 | Group B, SHP611 | Group C, SHP611 | Group F, SHP611 | GLIA-MLD Matched External Control for Group A
Started | 15 | 5 | 6 | 9 | 33 (Participants from GLIA-MLD study, part of GLIA-CTN study (NCT03047369).)
Completed | 12 | 3 | 5 | 9 | 0
Not Completed | 3 | 2 | 1 | 0 | 33
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by parent/guardian | 1 | 1 | 0 | 0 | 0
Not completed — Ongoing (Participants in GLIA-MLD, [part of GLIA-CTN study]) | 0 | 0 | 0 | 0 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A, SHP611 | Group B, SHP611 | Group C, SHP611 | Group F, SHP611 | GLIA-MLD Matched External Control for Group A | Total
Number analyzed (Participants) | 15 | 5 | 6 | 9 | 33 | 68
Age, Continuous [Mean (Standard Deviation); unit: months] | 18.27 (4.008) | 20.80 (4.658) | 17.67 (7.448) | 17.44 (4.746) | 14.76 (3.751) | 16.59 (4.692)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 2 | 4 | 15 | 36
  Male | 4 | 1 | 4 | 5 | 18 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 1 | 2 | 8
  Not Hispanic or Latino | 8 | 4 | 2 | 8 | 9 | 31
  Unknown or Not Reported | 4 | 0 | 3 | 0 | 22 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 2 | 0 | 0 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 1 | 3
  White | 12 | 5 | 5 | 7 | 13 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 17 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent Probability of Free of Loss of Locomotion in the Last Time Interval Up to 2 Years (Week 106) Based on GMFC-MLD for SHP611 Group A and GLIA-MLD Matched External Control
Description: Loss of locomotion was estimated using interval censoring survival analysis. Survival probability free of loss of locomotion based on GMFC-MLD was estimated up to Week 106 (or two years), with associated 2-sided 95 percent (%) confidence interval (CI).
  GMFC-MLD scale consists of 7 categories, scores ranging from 0 (walking without support with quality of performance normal for age) to 6 (loss of any locomotion as well as loss of any head and trunk control). Higher scores mean a worse outcome. The data was reported in terms of Mean as survival function was quantified using a weighted average of percentage of participants not reaching the event of interest, with weights derived from the relative size of treated and control units in the strata used for the stratified log-rank test in the primary analysis.
Time Frame: Baseline up to Week 106
Population: The modified full analysis set (mFAS) included all participants from Group A who received at least 1 dose of SHP611 and had at least a screening GMFC-MLD assessment, and the matched external control participants for Group A from GLIA-MLD natural history study. As per planned analysis, this outcome measure was assessed in Group A and GLIA-MLD matched external control for Group A.
Measure: Mean (95% Confidence Interval); unit: percent probability
Arm/Group | Group A, SHP611 | GLIA-MLD Matched External Control for Group A
Number analyzed (Participants) | 15 | 33
percent probability | 7.1 [0 to 20.2] | 9.4 [0 to 24.4]
Statistical Analysis 1: Comparison: Group A, SHP611 vs GLIA-MLD Matched External Control for Group A; Interval censoring survival analysis; Test type: Superiority — Survival probability free of loss of locomotion estimated up to Week 106 (or two years); p = 0.585, Log Rank — One-sided, over time intervals during entire follow-up. Stratified generalized log-rank test was used, where matching identification created from matching process in SAS PSMATCH Procedure used as strata; Difference in survival probability (%) = -2.2, 95% CI 2-sided [-22.2 to 17.7] — For the shared time interval up to Week 106 (or two years)

2. Secondary Outcome: Group A: Number of Participants Who Maintained Their Gross Motor Function Evaluated by Using the GMFC-MLD at Week 106 Compared With Matched External Control Group Data
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

3. Secondary Outcome: Number of Participants With Change From Baseline in Gross Motor Function Evaluated by Using the GMFC-MLD at Week 106
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline, Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

4. Secondary Outcome: Group A: Number of Participants With Decline From Baseline in GMFC-LMD of More Than 2 Categories
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline, Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

5. Secondary Outcome: Group A: Time to Decline From Baseline in GMFC-MLD of More Than 2 Categories
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline, Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Sulfatides Levels at Week 106
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline, Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

7. Secondary Outcome: Percent Change From Baseline in Cerebrospinal Fluid (CSF) Sulfatides Levels at Week 106
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline, Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

8. Secondary Outcome: Group A: Number of Participants With Maintenance of Gross Motor Function at Week 106 Using Gross Motor Function Measure 88 (GMFM-88) Total Score
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

9. Secondary Outcome: Time to Unreversed Decline From Baseline in GMFM-88 Total Score of Greater Than (>) 20 Points or Unreversed Decline to Less Than (<) 40 Points Whichever Occurs First
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline, Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

10. Secondary Outcome: Change From Baseline in GMFM-88 Total Score at Week 106
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline, Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

11. Secondary Outcome: Group A: Number of Participants With GMFM-88 Total Score Decrease of <= 20 Points From Baseline and a Total Score >=40 Points at Week 106
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline, Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

12. Secondary Outcome: Number of Participants With Change From Baseline in Expressive Language Evaluated by Using the Expressive Language Function Classification in Metachromatic Leukodystrophy (ELFC-MLD) Scale Categories at Week 106
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline, Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Event (TEAEs)
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: From start of study drug administration up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

14. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Values at Week 106
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

15. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination Findings at Week 106
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

16. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Values at Week 106
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

17. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Cerebrospinal Fluid (CSF) Laboratory Parameters at Week 106
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

18. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to SHP611
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

19. Secondary Outcome: Number of Participants With IDDD Implantations
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

20. Secondary Outcome: Number of Participants With Any IDDD Related Malfunctions
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

21. Secondary Outcome: IDDD Longevity as Assessed by Time to IDDD Failure
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

22. Secondary Outcome: Number of Participants With TEAE Related to IDDD and Surgical Procedure
Description: Data collection is ongoing and detailed reporting will be available after the study completion date.
Time Frame: Baseline up to Week 106
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Week 106
Description: SAS included all participants who received at least 1 dose of SHP611 or participants who underwent the IDDD implantation procedure. As per planned analysis GLIA-MLD Matched External Control for Group A was not a part of safety analysis, so data was not collected and analyzed.
Groups:
- Group A, SHP611: Participants aged 18 to 48 months with GMFC-MLD Category of 1 or 2 received SHP611 150 mg IT via IDDD or LP once weekly for 106 weeks in primary treatment period. Participants who completed primary treatment period will be continued treatment in extension period up to Week 210 or beyond, until their parents/guardians decided to discontinue treatment; the sponsor discontinued the study; the participant discontinued from the study due to medical or safety concerns; or the product became commercially available in the participant's country of residence, whichever came first.
Arm/Group | Group A, SHP611 | Group B, SHP611 | Group C, SHP611 | Group F, SHP611
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/5 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 14/15 | 4/5 | 5/6 | 9/9
Other Adverse Events (participants affected / at risk) | 15/15 | 5/5 | 6/6 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A, SHP611 (N=15) | Group B, SHP611 (N=5) | Group C, SHP611 (N=6) | Group F, SHP611 (N=9)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Bacterial test positive (Investigations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
CNS ventriculitis (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
CSF eosinophil count increased (Investigations) | 0 | 0 | 0 | 1
Central nervous system infection (Infections and infestations) | 1 | 0 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 2 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Device breakage (Product Issues) | 1 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 1 | 1
Device failure (Product Issues) | 4 | 0 | 0 | 1
Device leakage (Product Issues) | 1 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 2 | 1 | 0
Eating disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Encephalitis autoimmune (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 2 | 0 | 2 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Implant site oedema (General disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 0 | 0 | 0
Infusion related hypersensitivity reaction (Immune system disorders) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 2 | 0 | 0
Parainfluenzae viral bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Pleocytosis (Nervous system disorders) | 1 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 3
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Procedural failure (General disorders) | 1 | 0 | 0 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 4 | 1 | 2 | 4
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 3
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 3 | 1 | 4 | 5
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 2 | 0 | 3 | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Weight gain poor (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A, SHP611 (N=15) | Group B, SHP611 (N=5) | Group C, SHP611 (N=6) | Group F, SHP611 (N=9)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Adverse drug reaction (General disorders) | 1 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 2 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 2
Albumin CSF increased (Investigations) | 2 | 0 | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anisocoria (Eye disorders) | 0 | 0 | 1 | 0
Anticonvulsant drug level abnormal (Investigations) | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Areflexia (Nervous system disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial test (Investigations) | 1 | 0 | 1 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 1
Blood albumin increased (Investigations) | 2 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 2
Blood creatinine decreased (Investigations) | 0 | 0 | 1 | 1
Blood iron increased (Investigations) | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 2 | 0
Body temperature decreased (Investigations) | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 3 | 1 | 0 | 2
Bone demineralisation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Breathing-related sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Bruxism (Psychiatric disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 10 | 0 | 3 | 1
CSF eosinophil count increased (Investigations) | 1 | 0 | 0 | 0
CSF glucose decreased (Investigations) | 1 | 0 | 1 | 1
CSF monocyte count increased (Investigations) | 0 | 0 | 0 | 1
CSF mononuclear cell count increased (Investigations) | 1 | 0 | 0 | 0
CSF neutrophil count increased (Investigations) | 0 | 1 | 0 | 0
CSF protein increased (Investigations) | 7 | 1 | 3 | 6
CSF red blood cell count positive (Investigations) | 0 | 0 | 1 | 1
CSF test abnormal (Investigations) | 0 | 0 | 1 | 1
CSF white blood cell count increased (Investigations) | 4 | 1 | 2 | 2
Catheter site bruise (General disorders) | 0 | 0 | 0 | 1
Catheter site dermatitis (General disorders) | 0 | 0 | 1 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 2
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 1
Catheter site mass (General disorders) | 1 | 0 | 0 | 0
Catheter site swelling (General disorders) | 1 | 1 | 1 | 1
Cerebellar atrophy (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral atrophy (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrospinal fistula (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 2 | 0 | 0 | 3
Chalazion (Eye disorders) | 0 | 0 | 2 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Chorea (Nervous system disorders) | 1 | 0 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Complication associated with device (General disorders) | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 3 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 12 | 3 | 4 | 5
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0 | 0
Coronavirus test (Investigations) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1 | 5
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0
Crying (General disorders) | 0 | 0 | 0 | 1
Crystal urine present (Investigations) | 0 | 0 | 0 | 2
Culture positive (Investigations) | 1 | 0 | 0 | 0
Cyanosis (Vascular disorders) | 0 | 0 | 0 | 1
Decerebrate posture (Nervous system disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 1 | 1
Decreased eye contact (Psychiatric disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Demyelination (Nervous system disorders) | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Developmental delay (General disorders) | 1 | 0 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 1 | 0
Device kink (Product Issues) | 1 | 0 | 0 | 0
Device leakage (Product Issues) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 1 | 4
Discomfort (General disorders) | 1 | 1 | 0 | 0
Disorganised speech (Psychiatric disorders) | 1 | 0 | 0 | 0
Drooling (Nervous system disorders) | 2 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dumping syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 5 | 1 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dysstasia (Nervous system disorders) | 1 | 0 | 0 | 0
Dystonia (Nervous system disorders) | 4 | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0
Eating disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Electroencephalogram abnormal (Investigations) | 1 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Erythema of eyelid (Eye disorders) | 1 | 0 | 0 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 1 | 0
Eye movement disorder (Eye disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 1 | 4 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Food refusal (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fungal foot infection (Infections and infestations) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 1 | 0 | 0
Gait spastic (Nervous system disorders) | 0 | 0 | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Gallbladder enlargement (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 2 | 4
Gastroenteritis (Infections and infestations) | 5 | 1 | 4 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3 | 2 | 3
Gaze palsy (Eye disorders) | 1 | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Granuloma (General disorders) | 1 | 0 | 0 | 0
Haematocrit increased (Investigations) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 1 | 0
Haemoglobin increased (Investigations) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1
Heart rate decreased (Investigations) | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 1 | 1
Hepatic enzyme abnormal (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 1
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 2
Human bocavirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Hypertonia (Nervous system disorders) | 1 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Implant site oedema (General disorders) | 2 | 0 | 0 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incision site swelling (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Infantile spitting up (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 2
Infusion related hypersensitivity reaction (Immune system disorders) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 2 | 2 | 0 | 3
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 1 | 0 | 0 | 0
Laryngitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 2
Leukodystrophy (Congenital, familial and genetic disorders) | 1 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lordosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Medical device site granuloma (General disorders) | 0 | 1 | 0 | 0
Medical device site haemorrhage (General disorders) | 0 | 0 | 1 | 0
Medical device site infection (Infections and infestations) | 3 | 0 | 0 | 0
Medical device site irritation (General disorders) | 0 | 0 | 0 | 1
Medical device site swelling (General disorders) | 0 | 0 | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Mite allergy (Immune system disorders) | 1 | 0 | 0 | 0
Moaning (General disorders) | 0 | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0 | 0
Muscle enzyme increased (Investigations) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasticity (Nervous system disorders) | 11 | 3 | 2 | 6
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 1 | 0
Myopia (Eye disorders) | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 3 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Nitrite urine (Investigations) | 1 | 0 | 0 | 0
Nitrite urine present (Investigations) | 0 | 0 | 1 | 2
Nodule (General disorders) | 0 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 2
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Optic atrophy (Eye disorders) | 1 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 3 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0 | 1 | 3
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | 1
Pain (General disorders) | 2 | 1 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 2 | 0 | 2 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 1
Pleocytosis (Nervous system disorders) | 2 | 0 | 0 | 2
Plicated tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 2 | 4
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pre-existing condition improved (General disorders) | 0 | 1 | 0 | 0
Precocious puberty (Endocrine disorders) | 0 | 1 | 0 | 0
Procedural anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 8 | 1 | 1 | 4
Procedural vomiting (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Protein urine (Investigations) | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 1 | 0 | 0 | 3
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Pyrexia (General disorders) | 13 | 3 | 4 | 9
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Red blood cell count increased (Investigations) | 1 | 0 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 1
Regressive behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1
Regurgitation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 2
Restlessness (Psychiatric disorders) | 2 | 0 | 1 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retinal dystrophy (Eye disorders) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 0 | 3 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 3
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 3 | 3 | 3 | 3
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 1
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 2 | 1 | 2 | 4
Seizure cluster (Nervous system disorders) | 1 | 0 | 1 | 0
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sleep deficit (Nervous system disorders) | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 4 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 2 | 1
Specific gravity urine increased (Investigations) | 1 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Staring (Psychiatric disorders) | 1 | 1 | 0 | 0
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Strabismus (Eye disorders) | 0 | 1 | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 2 | 1 | 5
Urinary tract infection (Infections and infestations) | 4 | 1 | 0 | 3
Urine analysis abnormal (Investigations) | 1 | 0 | 0 | 1
Urine transitional cells present (Investigations) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vancomycin infusion reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 2 | 0 | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Viral rash (Infections and infestations) | 1 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 1 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Vitamin D decreased (Investigations) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 2 | 3 | 8
Weight decreased (Investigations) | 0 | 0 | 2 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Wound drainage (Surgical and medical procedures) | 0 | 0 | 0 | 1
Xanthochromia (Investigations) | 1 | 0 | 0 | 0
pH urine increased (Investigations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT03771898/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT03771898/SAP_001.pdf